CLINICAL TRIAL: NCT04429841
Title: Operative and Long Term Oncological Outcomes After D2 Versus D1 Gastrectomy of Operable Gastric Cancer
Brief Title: D2 Versus D1 Gastrectomy of Operable Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Assistant professor of Surgery, Alexandria University
Other Study IDs: 302764
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Gastric Cancer
Keywords: Operable Gastric Cancer; D2 Gastrectomy; D1 Gastrectomy; Operative Mortality & Morbidity; Oncological Outcomes
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D1 Gastrectomy: Patients are managed by radical gastrectomy with D1 lymphadenectomy
  Interventions: Procedure: Radical gastrectomy with D1 lymphadenectomy
- D2 Gastrectomy: Patients are managed by radical gastrectomy with D2 lymphadenectomy
  Interventions: Procedure: Radical gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Procedure: Radical gastrectomy with D1 lymphadenectomy
  Groups: D1 Gastrectomy
Procedure: Radical gastrectomy with D2 lymphadenectomy
  Groups: D2 Gastrectomy

SUMMARY:
Surgery is the mainstay treatment of operable gastric carcinoma but the optimal extent of lymph node (LN) dissection is controversial. The aim of this observational study is to assess the outcomes after curative D2 compared to D1 gastrectomy of operable gastric carcinoma regarding operative and long term oncological outcomes.

DETAILED DESCRIPTION:
This observational study included 80 consecutive patients presented by operable gastric cancer treated by D2 gastrectomy at Alexandria University hospital between January 2010 and January 2016, (Group I). Another 68 consecutive patients presented by operable gastric cancer treated by D1 gastrectomy earlier during the same period were included as a control (Group II). All patients had undergone preoperative gastroscopy and biopsy, chest and abdomen computed tomography (CT). All surgeries were performed by surgeons experienced in both D1 and D2 dissection and a standardized protocol for D1 and D2 gastrectomy was followed in all patients. The type of gastrectomy (distal or total) was done according to the site of the tumor; distal gastrectomy was done if there is a free safety margin of 4 cm beyond the proximal resection line otherwise total gastrectomy was done. Resection of the spleen and/or pancreatic tail were done if directly invaded by the primary tumor or metastatic LN. Patients with p T2 or greater, or with positive LN received adjuvant chemotherapy. Follow up was done as outpatient visits for average 5 years. Both groups were compared regarding postoperative morbidity and mortality, disease recurrence and survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 80 years with a histologically confirmed operable adenocarcinoma of the stomach with complete follow up after surgery for average 5 years

Exclusion Criteria:

* Complicated gastric cancer (obstructed or perforated)
* Irresectable or metastatic disease
* Previous or coexisting cancer
* Prior gastric surgery.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This observational study included 80 consecutive patients presented by operable gastric cancer treated by D2 gastrectomy at Alexandria University hospital between January 2010 and January 2016, (Group I). Another 68 consecutive patients presented by operable gastric cancer treated by D1 gastrectomy earlier during the same period were included as a control (Group II).
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity rate | 30 days after surgery
  Frequency of early postoperative complications
Operative mortality rate | 30 days after surgery
  Frequency of early postoperative mortality

SECONDARY OUTCOMES:
5 years Recurrence rate | 5 years after surgery
  Frequency of tumor recurrence within 5 years after curative surgery
5 years Cancer specific mortality rate | 5 years after surgery
  Frequency of Cancer specific mortality within 5 years after curative surgery
5 years Disease free survival rate | 5 years after surgery
  Percentage of patients survived for 5 years after surgery without tumor recurrence
5 years Overall survival rate | 5 years after surgery
  Percentage of patients survived for 5 years after surgery with/without tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmessiry, MD, Principal Investigator — Assistant Professor of Surgery
Locations (1):
- Alexandria, Egypt

REFERENCES:
- [Background] Tamura S, Takeno A, Miki H. Lymph node dissection in curative gastrectomy for advanced gastric cancer. Int J Surg Oncol. 2011;2011:748745. doi: 10.1155/2011/748745. Epub 2011 Jun 14. PMID 22312521
- [Background] Hartgrink HH, van de Velde CJ, Putter H, Bonenkamp JJ, Klein Kranenbarg E, Songun I, Welvaart K, van Krieken JH, Meijer S, Plukker JT, van Elk PJ, Obertop H, Gouma DJ, van Lanschot JJ, Taat CW, de Graaf PW, von Meyenfeldt MF, Tilanus H, Sasako M. Extended lymph node dissection for gastric cancer: who may benefit? Final results of the randomized Dutch gastric cancer group trial. J Clin Oncol. 2004 Jun 1;22(11):2069-77. doi: 10.1200/JCO.2004.08.026. Epub 2004 Apr 13. PMID 15082726